CLINICAL TRIAL: NCT02952703
Title: Disseminating and Implementing a Smoking Cessation Program Fro Pregnant and Postpartum Women
Brief Title: Disseminating and Implementing a Smoking Cessation Program for Pregnant and Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-1046
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Smoking; Tobacco Use Disorder
MeSH Terms: conditions — Smoking; Tobacco Use Disorder | interventions — Fertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Breath (Active Comparator): brief pre-natal smoking cessation counseling
  Interventions: Behavioral: brief pre-delivery smoking cessation counseling
- Striving to Quit (Experimental): Additional pre-natal counseling (in-person and telephonic); post delivery counseling (in-person and telephonic) and incentives
  Interventions: Behavioral: additional pre-delivery smoking cessation counseling; Behavioral: post- delivery smoking cessation counseling; Behavioral: incentives

INTERVENTIONS:
Behavioral: brief pre-delivery smoking cessation counseling
  Arms: First Breath
Behavioral: additional pre-delivery smoking cessation counseling
  Arms: Striving to Quit
Behavioral: post- delivery smoking cessation counseling
  Arms: Striving to Quit
Behavioral: incentives
  Arms: Striving to Quit

SUMMARY:
This study tests whether a smoking cessation intervention for pregnant women that extends postpartum (Striving to Quit (STQ)) can be implemented and disseminated outside of the research environment that established its effectiveness (40% maintained biochemically verified 6-month abstinence). The research aim is:

Is Striving to Quit more effective in achieving postpartum smoking cessation than "First Breath," the current standard of care for pregnant women in Wisconsin who smoke?

250 women will be randomized into one of two study groups. Pregnant women in Group A (n=125) will receive the existing First Breath prenatal intervention. Those in Group B (Striving to Quit (STQ), n=125) will receive all Group A interventions, plus 1 additional prenatal home visit, 3 postpartum in-home smoking cessation counseling visits, 3 postpartum phone calls, and up to an additional $100 in gift cards. The primary outcome will be biochemically confirmed smoking cessation at 6-months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant;
* enrolled in First Breath;
* Resides in Wisconsin counties of Calumet, Fond Du Lac, Kewaunee, Menominee, Oconto, Shawno, Sheyboygan, Winnebago, Door, Brown, Outagamie, Manitowac, or Waupaca;
* English speaking;
* willingness to quit or reduce smoking in next 30 days or if already quit, desire to remain quit after delivery;
* daily smoking (at least 1 cigarette/day for at least 1 week in past 6 months;
* willing to provide updates in contact information

Exclusion Criteria:

* not pregnant;
* not smoking in past 6 months;
* involved in another smoking research study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-11; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Biochemically verified smoking abstinence | 6 months post intervention
  Biochemically verified smoking abstinence: Breath Carbon Monoxide (CO)<9ppm

SECONDARY OUTCOMES:
Motivation to quit/remain quit | 6 months post intervention
  Motivation to quit/remain quit measured on a 5 point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT02952703/Prot_SAP_ICF_000.pdf